CLINICAL TRIAL: NCT04853485
Title: Repetitive Transcranial Magnetic Stimulation in Subjects With Early Psychosis and The Functional Connectivity Biotypes
Brief Title: Repetitive Transcranial Magnetic Stimulation in Early Psychosis and The Functional Connectivity Biotypes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Suzhou Psychiatric Hospital (Other); Guangzhou Psychiatric Hospital (Other Government); Shenzhen Kangning Hospital (Other); Tianjin Anding Hospital (Other); Nantong Fourth People's Hospital & Nantong Brain Hospital (Unknown)
Responsible Party: Principal Investigator, Jijun Wang, Professor of Department of Psychiatry, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRC2018ZD01
Record Dates: First submitted 2021-03-31; First posted 2021-04-21 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Schizophrenia; Psychosis; First Episode Psychosis; Clinical High Risk
Keywords: schizophrenia; prodromal phase; biotypes; target optimizing; precision calculation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Active TMS targeting both cerebellum and right dorsolateral prefrontal cortex. (Active Comparator): Subjects identified as with prominent negative symptoms will be randomized into active group, who will receive active rTMS over cerebellum and right dorsolateral prefrontal cortex navigated by individual MRI.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Sham TMS targeting both cerebellum and right dorsolateral prefrontal cortex (Sham Comparator): Subjects identified as with prominent negative symptoms will be randomized into sham group, who will receive sham rTMS over cerebellum and right dorsolateral prefrontal cortex navigated by individual MRI.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Active TMS targeting left inferior parietal lobule (Active Comparator): Subjects identified with prominent cognition deficits wil be randomized into active group, who will receive active rTMS over left inferior parietal lobule, navigated by individual MRI and functional connectivity map with left hippocampus.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Sham TMS targeting left inferior parietal lobule (Placebo Comparator): Subjects identified with prominent cognition deficits wil be randomized into sham group, who will receive sham rTMS over left inferior parietal lobule, navigated by individual MRI and functional connectivity map with left hippocampus.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Active deep TMS using Brainways H7 coil targeting ACC (Active Comparator): Subjects identified as with positive symptoms will be randomized into active group, who will receive active deep rTMS over ACC using H7 coil.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Sham deep TMS using Brainways H7 coil targeting ACC (Placebo Comparator): Subjects identified with positive symptoms will be randomized into sham group, who will receive sham deep rTMS over ACC using H7 coil.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — All subjects with early psychosis will be divided into three subgroups determined by their psychotic symptoms and cognition. There are three rTMS strategies: (1) For subgroup 1, characterized by negative symptoms, iTBS over cerebellum and 1 Hz over right DLPFC; (2) For subgroup 2, characterized by cognition deficits, 20 Hz over the left inferior parietal cortex; (3) For subgroup 3, characterized by positive symptoms: 10 Hz over ACC. Ten to twenty sessions of rTMS will be delivered to each patients during the intervention period.

SUMMARY:
The present study plans to explore different cortical targets of repetitive transcranial magnetic stimulation (rTMS) for populations at the early phase of psychosis, including those at clinical high risk of psychosis and in the first episode of psychosis. The clinical augmentation efficacy will be associated with the brain functional connectivity of these populations.

DETAILED DESCRIPTION:
Schizophrenia is a life long illness, the management of its early stage is the key in its long term outcomes. The early stage of schizophrenia includes the prodromal and first episode, during which the patients present psychotic symptoms (positive symptoms, negative symptoms) and cognition deficits. Antipsychotics are often prescribed to treat these symptoms, but more than one third patients do not respond well. Regarding cognition deficits, for example, while the visual spatial learning evaluated using Brief Visuospatial Memory Test-Revised (BVMT-R) of The Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) may play an important role in the conversion of psychosis in the prodromal phase, there is still no corresponding intervention.

Repetitive transcranial magnetic stimulation (rTMS) is a new non-invasive brain stimulation. In previous studies, its applications mainly focus on negative symptoms and demonstrate promising findings. However, its efficacy has much needing improvement, urgently needing target optimizing and precision, especially according to the prominent complaints of patients. To solve this issue, the present project proposed to make efforts in 3 aspects: to recruit patients in early phase of illness, to administer rTMS of different protocols according to the symptoms and cognition, and to associate the biotypes of functional connectivity with rTMS's efficacy. All subjects will receive MRI scan before rTMS intervention in the present study. The clinical efficacy of rTMS of the present protocol will be applied to validate the biotypes of functional connectivity in early psychosis. The biotypes will be determined using an existing independent dataset, which include 650 available cases of resting MRI (including 400 patients in prodromal phase, 100 patients with first episode and 150 controls).

Individual rTMS target will be optimized basing individual neuroimaging navigation. In the present protocol, we will recruit 300 new cases and perform a multicenter and randomized clinical trial to test the efficacy of our optimized rTMS protocols. All patients will be stratified according to their negative symptoms, positive symptom and cognition, and this will be determined by a panel of psychiatrists and rTMS therapists. It is estimated that about 100 cases in each of three subgroups. Subgroup 1 is characterized by prominent negative symptoms and will receives rTMS over cerebellum and right dorsolateral prefrontal cortex. Subgroup 2 is characterized by prominent cognition deficits and will receive rTMS over left inferior parietal lobule, navigated by individual MRI and functional connectivity map with left hippocampus. Subgroup 3 is characterized by positive symptoms and will receive deep rTMS over ACC using H7 coil. The present project, if being performed successfully, will promote the non-invasive physical therapy in psychiatry to a significantly higher level.

ELIGIBILITY:
For subjects at clinical high-risk for psychosis

Inclusion Criteria:

* Meeting the syndrome of clinical high risk of psychosis, identified by a face-to-face interview using the Chinese version of Structured Interview for Prodromal Syndromes / Scale of Prodromal Symptoms (SIPS/SOPS);
* Given the written consent for participation.
* Age between 14-45 years old;
* IQ>69;
* PANSS total scores >= 55 or BVMT-R score <= 26;

Exclusion Criteria:

* any contraindication to TMS treatment or magnetic resonance imaging (MRI)
* substance or alcohol abuse within recent three months
* any sensorimotor disorder (e.g., hearing disorder, lose one's sight), or any neurological disease (brain injury, epilepsy ) or any other physical disease which may lead to psychotic symptoms.

For subjects with first-episode schizophrenia

Inclusion Criteria:

* Meeting the DSM-V diagnostic criteria for schizophrenia spectrum disorders;
* Given the written consent for participation.
* Age between 14-45 years old;
* IQ>69;
* during the first episode without a full remission;
* PANSS total scores >= 55 or BVMT-R score <= 26;
* within receiving rTMS, patients can receive second-generation antipsychotics except clozapine with stable dosages

Exclusion Criteria:

* any contraindication to TMS treatment or magnetic resonance imaging (MRI)
* substance or alcohol abuse within recent three months
* any sensorimotor disorder (e.g., hearing disorder, lose one's sight), or any neurological disease (brain injury, epilepsy) or any other physical disease which may lead to psychotic symptoms.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate (the number of non-responders) for subgroup 1 and subgroup 3 | Within 24 hours after the rTMS intervention
  Response or responder will be determined by the reduction of PANSS total scores >= 25%
Improvement on cognition for subgroup 2 | Within 24 hours after the rTMS intervention
  Change in BVMT-R score as measured by MCCB

SECONDARY OUTCOMES:
Improvement of psychotic symptoms | Within 24 hours after the rTMS intervention
  The changes of PANSS scores and sub-scale scores
Improvement of prodromal symptoms | Within 24 hours after the rTMS intervention
  The changes of SOPS scores and sub-scale scores
Improvement of cognitive function | Within 24 hours after the rTMS intervention
  The changes of all cognitive domains assessed by MCCB
Improvement of global functioning | Within 24 hours after the rTMS intervention
  The GAF changes
Functional connectivity | Within 1week after the rTMS intervention
  changes of whole-brain functional connectivity patterns
side effect and safety | during and after rTMS intervention
  the frequency and severity of side effects
clinical outcome | 1 year
  remission, non-remission or relapse
The accuracy of prediction with functional connectivity biotypes at baseline | 1 year
  The association of clinical outcomes after rTMS intervention with functional connectivity biotypes at baseline
change in individualized psychosis risk score | Within 24 hours after the rTMS intervention
  For subjects at clinical high risk of psychosis, individualized psychosis risk score will be calculated using clinical symptoms and cognition, which indicate the psychosis risk in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Jijun Wang, M.D., Ph.D, Principal Investigator — Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine
Locations (6):
- China (6):
  - The Affiliated Brain Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Nantong Fourth People's Hospital & Nantong Brain Hospital, Nantong, Jiangsu
  - Suzhou Guangji Hospital, Suzhou, Jiangsu
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Shenzhen Kangning Hospital, Shenzhen
  - Tianjin Anding Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cui H, Giuliano AJ, Zhang T, Xu L, Wei Y, Tang Y, Qian Z, Stone LM, Li H, Whitfield-Gabrieli S, Niznikiewicz M, Keshavan MS, Shenton ME, Wang J, Stone WS. Cognitive dysfunction in a psychotropic medication-naive, clinical high-risk sample from the ShangHai-At-Risk-for-Psychosis (SHARP) study: Associations with clinical outcomes. Schizophr Res. 2020 Dec;226:138-146. doi: 10.1016/j.schres.2020.06.018. Epub 2020 Jul 18. PMID 32694037
- [Background] Wang J, Zhou Y, Gan H, Pang J, Li H, Wang J, Li C. Efficacy Towards Negative Symptoms and Safety of Repetitive Transcranial Magnetic Stimulation Treatment for Patients with Schizophrenia: A Systematic Review. Shanghai Arch Psychiatry. 2017 Apr 25;29(2):61-76. doi: 10.11919/j.issn.1002-0829.217024. PMID 28765677
- [Background] Zhuo K, Tang Y, Song Z, Wang Y, Wang J, Qian Z, Li H, Xiang Q, Chen T, Yang Z, Xu Y, Fan X, Wang J, Liu D. Repetitive transcranial magnetic stimulation as an adjunctive treatment for negative symptoms and cognitive impairment in patients with schizophrenia: a randomized, double-blind, sham-controlled trial. Neuropsychiatr Dis Treat. 2019 May 8;15:1141-1150. doi: 10.2147/NDT.S196086. eCollection 2019. PMID 31190822
- [Background] Brady RO Jr, Gonsalvez I, Lee I, Ongur D, Seidman LJ, Schmahmann JD, Eack SM, Keshavan MS, Pascual-Leone A, Halko MA. Cerebellar-Prefrontal Network Connectivity and Negative Symptoms in Schizophrenia. Am J Psychiatry. 2019 Jul 1;176(7):512-520. doi: 10.1176/appi.ajp.2018.18040429. Epub 2019 Jan 30. PMID 30696271
- [Background] Tang Y, Jiao X, Wang J, Zhu T, Zhou J, Qian Z, Zhang T, Cui H, Li H, Tang X, Xu L, Zhang L, Wei Y, Sheng J, Liu L, Wang J. Dynamic Functional Connectivity Within the Fronto-Limbic Network Induced by Intermittent Theta-Burst Stimulation: A Pilot Study. Front Neurosci. 2019 Sep 13;13:944. doi: 10.3389/fnins.2019.00944. eCollection 2019. PMID 31572111
- [Background] Tang Y, Xu L, Zhu T, Cui H, Qian Z, Kong G, Tang X, Wei Y, Zhang T, Hu Y, Sheng J, Wang J. Visuospatial Learning Selectively Enhanced by Personalized Transcranial Magnetic Stimulation over Parieto-Hippocampal Network among Patients at Clinical High-Risk for Psychosis. Schizophr Bull. 2023 Jul 4;49(4):923-932. doi: 10.1093/schbul/sbad015. PMID 36841956
- [Derived] Wang J, Wei Y, Hu Q, Tang Y, Zhu H, Wang J. The efficacy and safety of dual-target rTMS over dorsolateral prefrontal cortex (DLPFC) and cerebellum in the treatment of negative symptoms in first-episode schizophrenia: Protocol for a multicenter, randomized, double-blind, sham-controlled study. Schizophr Res Cogn. 2024 Nov 29;39:100339. doi: 10.1016/j.scog.2024.100339. eCollection 2025 Mar. PMID 39687049